CLINICAL TRIAL: NCT04852276
Title: Analysis of the Immune Response to COVID-19 Vaccination and Outcomes in Individuals With and Without Immune Deficiencies and Dysregulations
Brief Title: COVID-19 Vaccination and Outcomes in Individuals With and Without Immune Deficiencies and Dysregulations
Acronym: PERSIST
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000384; 000384-I (Other: NIAID)
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-10-06

CONDITIONS: Immunodeficiencies; Immune Dysregulations
Keywords: Adaptive immunity; clinical epidemiology; SARS-CoV-2; Coronavirus; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control participants: Control participants will be healthy volunteers, and may include unaffected relatives of immunodeficient/dysregulated participants
- Patients with immunodeficiencies and immune dysregulations: Affected patients with evidence of a primary or secondary immune deficiency or dysregulation

SUMMARY:
Background:

The immune system defends the body against disease and infection. Immune deficiencies are health conditions that decrease the strength of this response. Vaccines stimulate the immune system to create a defense against a specific type of germ. Researchers want to compare immune system responses to COVID-19 vaccines in people with and without immune deficiencies.

Objective:

To learn about how people with immune deficiencies respond to COVID-19 vaccines.

Eligibility:

People age 3 and older with an immune deficiency who plan to get a COVID-19 vaccine. Healthy volunteers are also needed.

Design:

Participants will be pre-screened for eligibility, including COVID-19 vaccination history and immune status.

Participants will give a blood sample before they get their first COVID-19 vaccine. Blood will be drawn from an arm vein using a needle. Blood can be drawn at the NIH, at a local doctor's office, or at a laboratory. It may also be drawn through a fingerstick at home. Participants will also complete 2 online surveys about their health and COVID-19 history. Additional surveys are optional.

Participants will give a second blood sample 2 to 4 weeks after they get the vaccine. They will complete 2 surveys about changes in their health and side effects from the vaccine.

If participants get another COVID-19 vaccine dose, they will repeat the blood draw and surveys 3 to 4 weeks later.

Participants may give 3 optional blood samples in the 24 months after their last vaccine. They may also give saliva samples every 2 weeks while they are in the study for 6 months following their last vaccine.

Participation will last from 1 month to 2 years after the participant's last vaccine.

DETAILED DESCRIPTION:
Study Description:

This prospective cohort study will assess the pre- and post-vaccination immune responses in individuals with select immunodeficiencies and immune dysregulations compared to healthy volunteers who receive a coronavirus disease 2019 (COVID-19) vaccine, as well as any adverse events (AEs) experienced after vaccination. All required study visits for this protocol may be conducted remotely; in-person visits at the NIH are optional. Subjects who have not yet been vaccinated will undergo baseline blood sampling using finger stick microsampler kits and/or venous blood draw within 7 days prior to receiving the vaccine. Additional samples will be requested from participants approximately 14-21 days after dose 1 and 21-28 days after dose 2 (if applicable). Optional samples may be collected at 6, 12, and 24 months post-vaccination. If subsequent booster doses are received while a participant is still on study, blood samples will again be requested approximately 28 days after each booster dose, through the 5th COVID-19 vaccine dose received, and then participants may proceed with the optional 6-, 12-, and 24-month follow-up sample collection. Participants who are able to attend in-person visits at NIH will have optional on-site blood draws 1 and 3 days after doses 1 and 2 (as applicable). Research evaluations will include baseline severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) antibody titers to the spike (S), nucleocapsid (N), and receptor binding domain (RBD) proteins, to assess pre-vaccination SARS-CoV-2 exposure and evaluate responses to vaccination. Additional immune markers of interest may include presence of autoantibodies, transcriptomic profiling, T-cell receptor (TCR) repertoire, among others. Participants who only submit finger stick home microsampler kits at the timepoints listed above will be evaluated for SARS-CoV-2 antibody titers and autoantibodies only. All subjects will be asked at baseline about prior COVID-19 diagnosis, symptoms, and severity, and will be asked additional questions at follow-up timepoints (including after additional booster doses) about vaccine AEs using standardized questionnaires.

Primary Objective:

To characterize the immune response to COVID-19 vaccination among immunodeficient and immune dysregulated individuals compared to healthy volunteers.

Secondary Objectives:

To characterize the COVID-19 vaccine-associated AEs among immunodeficient and immune dysregulated individuals compared to healthy volunteers.

Exploratory Objectives:

Assess the relationship between prior SARS-CoV-2 infection and vaccine-induced immune response.

To characterize pre-vaccine COVID-19 disease prevalence and severity among immunodeficient and immune dysregulated individuals.

To assess induction, strength, and durability of T- and B-cell specific immune responses to SARS-CoV-2 (as measured by frequency and diversity of SARS-CoV-2 specific T and B cell clonotypes and titers of specific antibody responses), and their correlation to the underlying immune deficiency/dysregulation.

To characterize auto-antibodies present in immunodeficient and immune dysregulated individuals before and after COVID-19 vaccination.

To assess the incidence of post-vaccination breakthrough SARS-CoV-2 infection and to determine the SARS-CoV-2 virus genomic sequence in such cases.

Primary Endpoint:

Change in S and RBD immunoglobulin G (IgG) antibody titer from baseline to 14-21 days or 21-28 days (depending on vaccine manufacturer and platform) after vaccine dose 1, and 21-28 days after dose 2 and any subsequent doses (depending on vaccine manufacturer and platform).

Secondary Endpoints:

Incidence of vaccine-associated AEs experienced by immunodeficient individuals compared to healthy volunteers.

Exploratory Endpoints:

Characterization of post-vaccine immune response and AEs in patients with antibody evidence of prior SARS-CoV-2 infection

Pre- and post-vaccination incidence of COVID-19-associated symptoms experienced in individuals with immune deficiency/dysregulation who are positive for SARS-CoV-2 by serology or diagnostic polymerase chain reaction (PCR).

Characterize how various forms of immune deficiency or dysregulation impact generation, strength, and durability of T- and B-cell responses.

Incidence of autoantibodies pre- and post-COVID-19 vaccination comparing individuals with immune deficiency/dysregulation to healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet the following criteria:

1. Aged 3 years and older.
2. Must be eligible to receive (based on official FDA authorization or approval) and scheduled to receive or have already received a COVID-19 vaccine outside of this facility.
3. Must meet the definition of affected participant or control participant:

   1. Affected participants must have evidence of a primary or secondary immune deficiency or dysregulation under another NIAID protocol or as documented by an outside physician.
   2. Control participants are healthy volunteers that do not have evidence of a primary or secondary immune deficiency or dysregulation and may include unaffected relatives of affected participants.
4. Ability to provide informed consent.
5. Willing to have blood samples stored for future research.
6. Able to proficiently speak, read, and write English.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Receipt of any other vaccine within 14 days prior to screening.
2. Planned non-COVID-19 vaccination within 28 days after COVID-19 vaccination(s).
3. Any condition that, in the opinion of the investigator, contraindicates participation in this study (e.g. specific autoinflammatory diseases, interferonopathies).
4. Self-reported history of HIV.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Immunodeficient individuals will be recruited from NIAID protocols that evaluate primary or secondary immune deficiencies. Potential subjects will be identified by discussion between the study teams and review of medical and research records if necessary. They may also be referred from community practitioners who see this population.Healthy adult volunteers will be recruited through the NIH Clinical Research Volunteer Program, the Office of Patient Recruitment, MMG Patient Recruitment, ResearchMatch, or BuildClinical. Volunteers will also be recruited from existing NIH protocols. Healthy relatives of immunodeficient participants can be recruited for participation as controls if they meet enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Ricotta, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szczawinska-Poplonyk A, Breborowicz A, Samara H, Ossowska L, Dworacki G. Impaired Antigen-Specific Immune Response to Vaccines in Children with Antibody Production Defects. Clin Vaccine Immunol. 2015 Aug;22(8):875-82. doi: 10.1128/CVI.00148-15. Epub 2015 May 27. PMID 26018535
- [Background] Bonilla FA. Vaccines in Patients with Primary Immune Deficiency. Immunol Allergy Clin North Am. 2020 Aug;40(3):421-435. doi: 10.1016/j.iac.2020.03.004. PMID 32654690
- [Background] Jackson LA, Anderson EJ, Rouphael NG, Roberts PC, Makhene M, Coler RN, McCullough MP, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott A, Flach B, Doria-Rose NA, Corbett KS, Morabito KM, O'Dell S, Schmidt SD, Swanson PA 2nd, Padilla M, Mascola JR, Neuzil KM, Bennett H, Sun W, Peters E, Makowski M, Albert J, Cross K, Buchanan W, Pikaart-Tautges R, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020 Nov 12;383(20):1920-1931. doi: 10.1056/NEJMoa2022483. Epub 2020 Jul 14. PMID 32663912
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000384-I.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2021 through December 2022. Immune deficient individuals were recruited from NIAID protocols evaluating immune deficiencies, referred from physicians, or self-referred. Healthy adult volunteers were recruited through various avenues. Healthy relatives of immunodeficient participants were recruited for participation as controls if they met enrollment criteria.
Groups:
- Immune Deficient/Disordered: Immune Deficient/Disordered participants must have evidence of a primary or secondary immune deficiency or dysregulation under another NIAID protocol or as documented by an outside physician.
- Healthy Control: Healthy volunteers do not have evidence of a primary or secondary immune deficiency or dysregulation and may include unaffected relatives of affected participants.
Period: Overall Study
Arm/Group | Immune Deficient/Disordered | Healthy Control
Started | 235 | 73
Completed | 192 | 58
Not Completed | 43 | 15
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 15 | 9
Not completed — Withdrawal by Subject | 26 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immune Deficient/Disordered | Healthy Control | Total
Number analyzed (Participants) | 235 | 73 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 7 | 38
  Between 18 and 65 years | 172 | 55 | 227
  >=65 years | 32 | 11 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (19) | 42 (19) | 43 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 45 | 190
  Male | 90 | 28 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 20
  Not Hispanic or Latino | 212 | 62 | 274
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 7 | 17
  White | 204 | 51 | 255
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 233 | 73 | 306
  Canada | 2 | 0 | 2
Antibody deficiency [Count of Participants; unit: Participants] | 54 | 0 | 54
Primary immune regulatory disorder [Count of Participants; unit: Participants] | 56 | 0 | 56
Combined immunodeficiency [Count of Participants; unit: Participants] | 13 | 0 | 13
Other inborn error of immunity [Count of Participants; unit: Participants] | 42 | 0 | 42
Other immune disorder [Count of Participants; unit: Participants] | 70 | 0 | 70
Healthy volunteer [Count of Participants; unit: Participants] | 0 | 73 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in S and Receptor Binding Domain (RBD) Immunoglobulin G (IgG) Antibody Titer From Baseline Depending on Vaccine Manufacturer and Platform
Description: To characterize the immune response to coronavirus disease 2019 (COVID-19) vaccination among immunodeficient and immune dysregulated individuals compared to healthy volunteers
Time Frame: Baseline, post dose 1 (14-21 days), and post dose 2 (21-28 days), depending on vaccine manufacturer and platform
Population: Analysis for these endpoints consisted only of participants who were enrolled and had provided samples at baseline and post-dose 1 or post-dose 1 and post-dose 2.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Immune Deficient/Disordered | Healthy Control
Number analyzed (Participants) | 95 | 27
ug/ml
  Change in anti-S titer from Baseline to Post-dose 1: number analyzed (Participants) | 43 | 10
  Change in anti-S titer from Baseline to Post-dose 1 | 0.447333 (1.118685) | 2.10678 (4.048595)
  Change in anti-S titer from Post-dose 1 to Post-dose 2: number analyzed (Participants) | 52 | 17
  Change in anti-S titer from Post-dose 1 to Post-dose 2 | 0.83819 (8.953689) | 2.8153 (5.749115)

2. Secondary Outcome: Incidence of Vaccine-associated Adverse Events (AE) Experienced by Immunodeficient Individuals Compared to Healthy Volunteers
Description: To characterize the COVID-19 vaccine-associated adverse events among immunodeficient and immune dysregulated individuals compared to healthy volunteers.
  Note on terminology: "No vaccine-associated side effects" means participants reported zero symptoms or reactions after vaccination. A "mild vaccine-associated side effect" means a participant reported any symptom/reaction and reported is as "mild" on the scale of "mild", "moderate", or "severe". A participant could have reported several mild symptom/reactions and several moderate or severe symptoms/reactions. Therefore, the number of mild, moderate, and severe vaccine-associated side effects will not sum to the total number of surveys completed.
Time Frame: Baseline up to a maximum of 24 months
Population: Analysis consisted of participants who returned each relevant survey on vaccine-associated events.
Measure: Number; unit: participants
Arm/Group | Immune Deficient/Disordered | Healthy Control
Number analyzed (Participants) | 212 | 60
participants
  Vaccine-associated side-effects after dose 1 : No vaccine-associated side effects: number analyzed (Participants) | 187 | 57
  Vaccine-associated side-effects after dose 1 : No vaccine-associated side effects | 31 | 6
  Vaccine-associated side-effects after dose 1 : Mild vaccine-associated side effects | 134 | 45
  Vaccine-associated side-effects after dose 1 : Moderate vaccine-associated side effects | 85 | 26
  Vaccine-associated side-effects after dose 1 : Severe vaccine-associated side effects | 19 | 9
  Vaccine-associated side-effects after dose 1 : Total Volunteers completing dose survey | 187 | 57
  Vaccine-associated side-effects after dose 2 : No vaccine-associated side effects: number analyzed (Participants) | 189 | 53
  Vaccine-associated side-effects after dose 2 : No vaccine-associated side effects | 28 | 8
  Vaccine-associated side-effects after dose 2 : Mild vaccine-associated side effects | 143 | 43
  Vaccine-associated side-effects after dose 2 : Moderate vaccine-associated side effects | 88 | 24
  Vaccine-associated side-effects after dose 2 : Severe vaccine-associated side effects | 16 | 6
  Vaccine-associated side-effects after dose 2 : Total Volunteers completing dose survey | 189 | 53
  Vaccine-associated side-effects after dose 3 : No vaccine-associated side effects: number analyzed (Participants) | 148 | 29
  Vaccine-associated side-effects after dose 3 : No vaccine-associated side effects | 16 | 7
  Vaccine-associated side-effects after dose 3 : Mild vaccine-associated side effects | 120 | 22
  Vaccine-associated side-effects after dose 3 : Moderate vaccine-associated side effects | 55 | 9
  Vaccine-associated side-effects after dose 3 : Severe vaccine-associated side effects | 19 | 1
  Vaccine-associated side-effects after dose 3 : Total Volunteers completing dose survey | 148 | 29
  Vaccine-associated side-effects after dose 4 : No vaccine-associated side effects: number analyzed (Participants) | 60 | 6
  Vaccine-associated side-effects after dose 4 : No vaccine-associated side effects | 7 | 0
  Vaccine-associated side-effects after dose 4 : Mild vaccine-associated side effects | 44 | 6
  Vaccine-associated side-effects after dose 4 : Moderate vaccine-associated side effects | 18 | 1
  Vaccine-associated side-effects after dose 4 : Severe vaccine-associated side effects | 3 | 0
  Vaccine-associated side-effects after dose 4 : Total Volunteers completing dose survey | 60 | 6
  Vaccine-associated side-effects after dose 5 : Mild vaccine-associated side effects | 4 | 0
  Vaccine-associated side-effects after dose 5 : Moderate vaccine-associated side effects | 1 | 0
  Vaccine-associated side-effects after dose 5 : Severe vaccine-associated side effects | 1 | 0
  Vaccine-associated side-effects after dose 5 : Total Volunteers completing dose survey | 4 | 0

ADVERSE EVENTS:
Time Frame: 2 years 4 months
Description: Serious and other (non-serious) adverse events were not collected or assessed as part of this study. This is an observational study, so no adverse events were monitored or assessed. Two participants died while on the study but that was purely observational and noted for our records, but had nothing to do with the study.
Arm/Group | Immune Deficient/Disordered | Healthy Control
All-Cause Mortality (participants affected / at risk) | 2/235 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a longitudinal observational study; participants could enroll at any point in their vaccine history. While 1 month post-vaccination samples were mandatory, subsequent samples were optional. Vaccination date and information was self-reported and sometimes resulted in delayed sample collection. Medical history, treatment status, and vaccine-associated side effects were self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT04852276/Prot_SAP_000.pdf
  • Informed Consent Form: Study Informed Consent (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT04852276/ICF_001.pdf
  • Informed Consent Form: Study Informed Consent (Assent Version) (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04852276/ICF_002.pdf